CLINICAL TRIAL: NCT00937950
Title: Gynaecological Follow-up of a Subset of 580299/008 Study Subjects
Brief Title: Gynaecological Follow-up of a Subset of 580299/008 (NCT00122681) Study Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112024; 2008-008124-33 (EudraCT Number)
Record Dates: First submitted 2009-07-02; First posted 2009-07-13 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; Papillomavirus; Human papillomavirus; Cervical cancer; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

ARMS (1):
- HPV-052 study subjects Group (Other): The study group consisted of a subset of HPV-008 (NCT00122681) study subjects (15-25 years old at first study vaccination), who at their last study visit (Visit 10, Month 48) in HPV-008 (NCT00122681) study displayed normal cervical cytology, but were tested positive for oncogenic HPV infection, or were pregnant and hence no cervical sample could be collected at their HPV-008 (NCT00122681) concluding visit.
  Interventions: Other: Gynaecological follow-up

INTERVENTIONS:
Other: Gynaecological follow-up — Subjects received a gynaecological follow-up with cytology and oncogenic HPV DNA testing every 12 months, for up to four years in this gynaecological follow-up study (HPV-052 EXT 008). No vaccine was administered in this extension study. Subjects received 3 doses of Cervarix/Havrix vaccine, administered intramuscularly, according to a 0, 1, 6-month vaccination schedule in the HPV-008 (NCT00122681) primary study.

SUMMARY:
This study is designed to provide up to four years of annual oncogenic HPV DNA testing and cervical cytology examination for NCT00122681 study subjects who displayed normal cervical cytology but tested positive for oncogenic HPV infection at their last NCT00122681 study visit (Visit 10, Month 48).

This follow-up study will also be offered to subjects who were pregnant at their last NCT00122681 study visit (Visit 10, Month 48) so that no cervical sample could be collected at that visit.

The objectives & outcome measures of the primary phase (study 008/580299) are presented in a separate protocol posting (NCT00122681).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to enrolment.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A subject previously enrolled in the study NCT00122681 and who fulfils either of the following criteria:

  * displayed normal cervical cytology but tested positive for oncogenic HPV infection at her last NCT00122681 study visit (Visit 10, Month 48).

or

- was pregnant at her last visit of the NCT00122681 study (Visit 10, Month 48) so that no cervical sample could be collected at that visit.

Exclusion Criteria:

* A subject who displayed normal cervical cytology and who was negative for oncogenic HPV infection at her last NCT00122681 study visit (Visit 10, Month 48).
* A subject who had a cervical lesion at her last NCT00122681 study visit (Visit 10, Month 48) or who had a cervical lesion that required treatment at the NCT00122681 exit colposcopy.
* A subject for whom the cervical cytology results from the last NCT00122681 study visit (Visit 10, Month 48) were unavailable for reasons other than pregnancy.

If at the time of enrolment the subject experiences heavy bleeding (menstruation or other) or heavy vaginal discharge, or is pregnant, the pelvic exam cannot be performed. The subject's first study visit will be deferred until condition is resolved according to investigator's medical judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2022 (Actual)
Dates: Start 2009-08-05 (Actual); Primary Completion 2014-01-20 (Actual); Study Completion 2014-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (76):
- United States (17):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pleasant Hills, Pennsylvania
  - GSK Investigational Site, Wenatchee, Washington
- Australia (5):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
- Brazil (3):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Curitiba
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Beauport, Quebec
  - GSK Investigational Site, Montreal, Quebec
- Finland (15):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kouvola
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Mikkeli
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Rauma
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vaasa
- Germany (12):
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Ravensburg, Baden-Wurttemberg
  - GSK Investigational Site, Rheinstetten, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Nordhausen, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Modena, Emilia-Romagna, Italy
- Philippines (6):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Laguna
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Los Banos, Laguna
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Manila
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (3):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 2022 subjects enrolled in this study, 19 were excluded for reasons of non-eligibility, hence only 2003 started the study.
Period: Overall Study
Arm/Group | HPV-052 Study Subjects Group
Started | 2003
Completed | 1787
Not Completed | 216
Not completed — Withdrawal by Subject | 23
Not completed — Migrated/moved from study area | 27
Not completed — Lost to Follow-up | 144
Not completed — Missing confirmed | 4
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 2003
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.3 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2003
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 58
  Race: White/Caucasian | 1211
  Race: Arabic/north African | 4
  Race: East & south east Asian | 549
  Race: South Asian | 3
  Race: Hispanic | 21
  Race: Chinese | 106
  Race: Indian | 1
  Race: Not specified | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With HPV DNA in Cervical Samples by Hybrid Capture 2 Test (HCII)
Description: Subjects who presented oncogenic HPV DNA in cervical samples by HPV DNA testing. The presence of oncogenic HPV infection was determined by the Hybrid Capture 2 (HCII) test, which detects HPV DNA types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 and 68.
  Missing = For some of the subjects whose result was indicated as quantity not sufficient (QNS).
Time Frame: At Months 12, 24, 36, 48
Population: The analysis was based on the Total HPV-052 cohort, which included subjects with available data at the considered time points and who at their last HPV-008 (NCT00122681) study visit displayed normal cervical cytology but tested positive for oncogenic HPV infection or were pregnant so that no cervical sample could be collected at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 1467
Participants
  Positive DNA (Month 12 Post HPV-008) | 615
  Negative DNA (Month 12 Post HPV-008) | 828
  Missing DNA (Month 12 Post HPV-008) | 24
  Positive DNA (Month 24 Post HPV-008): number analyzed (Participants) | 869
  Positive DNA (Month 24 Post HPV-008) | 418
  Negative DNA (Month 24 Post HPV-008): number analyzed (Participants) | 869
  Negative DNA (Month 24 Post HPV-008) | 444
  Missing DNA (Month 24 Post HPV-008): number analyzed (Participants) | 869
  Missing DNA (Month 24 Post HPV-008) | 7
  Positive DNA (Month 36 Post HPV-008): number analyzed (Participants) | 495
  Positive DNA (Month 36 Post HPV-008) | 255
  Negative DNA (Month 36 Post HPV-008): number analyzed (Participants) | 495
  Negative DNA (Month 36 Post HPV-008) | 236
  Missing DNA (Month 36 Post HPV-008): number analyzed (Participants) | 495
  Missing DNA (Month 36 Post HPV-008) | 4
  Positive DNA (Month 48 Post HPV-008): number analyzed (Participants) | 258
  Positive DNA (Month 48 Post HPV-008) | 144
  Negative DNA (Month 48 Post HPV-008): number analyzed (Participants) | 258
  Negative DNA (Month 48 Post HPV-008) | 107
  Missing DNA (Month 48 Post HPV-008): number analyzed (Participants) | 258
  Missing DNA (Month 48 Post HPV-008) | 7

2. Primary Outcome: Number of Subjects With Colposcopy Referral and Colposcopy Adequacy
Description: Subjects with normal cervical cytology, who were found to be oncogenic HPV DNA positive in two subsequent tests, were referred to colposcopy. The result of the subjects' last HPV-008 study visit was taken into account at Visit 1. Subjects with a single cervical cytology reading of ≥ atypical squamous cells of undetermined significance (ASC-US) positive for oncogenic HPV DNA were referred for colposcopy. Subjects with a single cervical cytology reading of ≥ low grade squamous intraepithelial lesion (LSIL) were referred to colposcopy, irrespective of their oncogenic HPV DNA test result.
Time Frame: At Months 12, 24, 36, 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 2003
Participants
  Colposcopy referral (Month 12) Yes | 572
  Colposcopy referral (Month 12) No | 1429
  Colposcopy referral (Month 12) Missing | 2
  Algorithm respected (Month 12) Yes: number analyzed (Participants) | 392
  Algorithm respected (Month 12) Yes | 371
  Algorithm respected (Month 12) No: number analyzed (Participants) | 392
  Algorithm respected (Month 12) No | 21
  Colposcopy adequacy (Month12),Satisfactory: number analyzed (Participants) | 392
  Colposcopy adequacy (Month12),Satisfactory | 370
  Colposcopy adequacy (Month12), Unsatisfactory: number analyzed (Participants) | 392
  Colposcopy adequacy (Month12), Unsatisfactory | 18
  Colposcopy adequacy (Month 12), Missing: number analyzed (Participants) | 392
  Colposcopy adequacy (Month 12), Missing | 4
  Colposcopy referral (Month 24) Yes | 385
  Colposcopy referral (Month 24) No | 1615
  Colposcopy referral (Month 24) Missing | 3
  Algorithm respected (Month 24) Yes: number analyzed (Participants) | 263
  Algorithm respected (Month 24) Yes | 254
  Algorithm respected (Month 24) No: number analyzed (Participants) | 263
  Algorithm respected (Month 24) No | 8
  Algorithm respected (Month 24) Missing: number analyzed (Participants) | 263
  Algorithm respected (Month 24) Missing | 1
  Colposcopy adequacy (Month24), Satisfactory: number analyzed (Participants) | 263
  Colposcopy adequacy (Month24), Satisfactory | 245
  Colposcopy adequacy(Month24),Unsatisfactory: number analyzed (Participants) | 263
  Colposcopy adequacy(Month24),Unsatisfactory | 14
  Colposcopy adequacy (Month 24), Missing: number analyzed (Participants) | 263
  Colposcopy adequacy (Month 24), Missing | 4
  Colposcopy referral (Month 36) Yes | 224
  Colposcopy referral (Month 36) No | 1776
  Colposcopy referral (Month 36) Missing | 3
  Algorithm respected (Month 36) Yes: number analyzed (Participants) | 158
  Algorithm respected (Month 36) Yes | 154
  Algorithm respected (Month 36) No: number analyzed (Participants) | 158
  Algorithm respected (Month 36) No | 4
  Colposcopy adequacy (Month36), Satisfactory: number analyzed (Participants) | 158
  Colposcopy adequacy (Month36), Satisfactory | 150
  Colposcopy adequacy(Month36), Unsatisfactory: number analyzed (Participants) | 158
  Colposcopy adequacy(Month36), Unsatisfactory | 7
  Colposcopy adequacy (Month 36), Missing: number analyzed (Participants) | 158
  Colposcopy adequacy (Month 36), Missing | 1
  Colposcopy referral (Month 48) Yes | 133
  Colposcopy referral (Month 48) No | 1867
  Colposcopy referral (Month 48) Missing | 3
  Algorithm respected (Month 48) Yes: number analyzed (Participants) | 96
  Algorithm respected (Month 48) Yes | 96
  Algorithm respected (Month 48) No: number analyzed (Participants) | 96
  Algorithm respected (Month 48) No | 0
  Colposcopy adequacy (Month48), Satisfactory: number analyzed (Participants) | 96
  Colposcopy adequacy (Month48), Satisfactory | 92
  Colposcopy adequacy (Month48), Unsatisfactory: number analyzed (Participants) | 96
  Colposcopy adequacy (Month48), Unsatisfactory | 3
  Colposcopy adequacy (Month 48), Missing: number analyzed (Participants) | 96
  Colposcopy adequacy (Month 48), Missing | 1

3. Primary Outcome: Number of Subjects With Cytological Abnormalities in Cervical Samples by ThinPrep PapTest
Description: Subjects who presented normal, ASC-US (Atypical Squamous Cell of Undetermined Significance), LSIL (Low-grade Squamous Intraepithelial Lesions), HSIL (High-grade Squamous Intraepithelial Lesions), AGC (Atypical Glandular Cells), ASC-H (Atypical Squamous Cells cannot exclude HSIL) cervical cytology.
  Cervical cytology examination was performed using the ThinPrep PapTest. Note: One subject may have presented with different cytology results at the yearly visit throughout the maximum 4-year follow-up period and therefore may be counted in more than one result category in the analysis.
Time Frame: At Months 12, 24, 36, 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 1467
Participants
  Normal, Month 12 | 1193
  ASC-US, Month 12 | 154
  ASC-H, Month 12 | 8
  LSIL, Month 12 | 100
  HSIL, Month 12 | 8
  AGC, Month 12 | 4
  Normal, Month 24: number analyzed (Participants) | 867
  Normal, Month 24 | 662
  ASC-US, Month 24: number analyzed (Participants) | 867
  ASC-US, Month 24 | 117
  ASC-H, Month 24: number analyzed (Participants) | 867
  ASC-H, Month 24 | 11
  LSIL, Month 24: number analyzed (Participants) | 867
  LSIL, Month 24 | 68
  HSIL, Month 24: number analyzed (Participants) | 867
  HSIL, Month 24 | 7
  AGC, Month 24: number analyzed (Participants) | 867
  AGC, Month 24 | 2
  Normal, Month 36: number analyzed (Participants) | 494
  Normal, Month 36 | 390
  ASC-US, Month 36: number analyzed (Participants) | 494
  ASC-US, Month 36 | 58
  ASC-H, Month 36: number analyzed (Participants) | 494
  ASC-H, Month 36 | 4
  LSIL, Month 36: number analyzed (Participants) | 494
  LSIL, Month 36 | 34
  HSIL, Month 36: number analyzed (Participants) | 494
  HSIL, Month 36 | 5
  AGC, Month 36: number analyzed (Participants) | 494
  AGC, Month 36 | 3
  Normal, Month 48: number analyzed (Participants) | 258
  Normal, Month 48 | 206
  ASC-US, Month 48: number analyzed (Participants) | 258
  ASC-US, Month 48 | 28
  ASC-H, Month 48: number analyzed (Participants) | 258
  ASC-H, Month 48 | 0
  LSIL, Month 48: number analyzed (Participants) | 258
  LSIL, Month 48 | 16
  HSIL, Month 48: number analyzed (Participants) | 258
  HSIL, Month 48 | 6
  AGC, Month 48: number analyzed (Participants) | 258
  AGC, Month 48 | 2

4. Primary Outcome: Number of Subjects With Cervical Biopsy Results at Month 12
Description: Subjects with negative and positive cervical biopsy results for only CIN1, only CIN2, only CIN3, CIN1 and CIN2, CIN1 and CIN3, CIN2 and CIN3, CIN1 and CIN2 and CIN3, AIS, Invasive malignancy, other.
  CIN = Cervical intraepithelial neoplasia. CIN1/CIN2/CIN3 = Cervical intraepithelial neoplasia grade 1/grade 2/grade 3.
  Note: Only CIN1/Only CIN2/Only CIN3 categories contain the subject who has only CIN1/CIN2/CIN3, but not the combinations.
Time Frame: At Month 12
Population: The analysis was based on the Total HPV-052 cohort, which included subjects for whom data were available at the considered time point and who at their last HPV-008 (NCT00122681) study visit displayed normal cervical cytology but tested positive for oncogenic HPV infection or were pregnant so that no cervical sample could be collected at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 199
Participants
  Negative | 76
  Only CIN1(positive) | 41
  Only CIN1(negative) | 158
  Only CIN2 (positive) | 18
  Only CIN2 (negative) | 181
  Only CIN3 (positive) | 8
  Only CIN3 (negative) | 191
  CIN1 and CIN2 (positive) | 3
  CIN1 and CIN2(negative) | 196
  CIN1 and CIN3(positive) | 1
  CIN1 and CIN3 (negative) | 198
  CIN2 and CIN3 (positive) | 1
  CIN2 and CIN3 (negative) | 198
  CIN1 and CIN2 and CIN3 (positive) | 0
  CIN1 and CIN2 and CIN3 (negative) | 199
  AIS (positive) | 0
  AIS (negative) | 199
  Invasive malignancy (positive) | 0
  Invasive malignancy (negative) | 199
  Other | 85

5. Primary Outcome: Number of Subjects With Cervical Biopsy Results at Month 24
Description: as for outcome 4
Time Frame: At Month 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 147
Participants
  Negative | 38
  Only CIN1(positive) | 47
  Only CIN1(negative) | 100
  Only CIN2 (positive) | 8
  Only CIN2 (negative) | 139
  Only CIN3 (positive) | 8
  Only CIN3 (negative) | 139
  CIN1 and CIN2 (positive) | 2
  CIN1 and CIN2(negative) | 145
  CIN1 and CIN3(positive) | 0
  CIN1 and CIN3 (negative) | 147
  CIN2 and CIN3 (positive) | 1
  CIN2 and CIN3 (negative) | 146
  CIN1 and CIN2 and CIN3 (positive) | 0
  CIN1 and CIN2 and CIN3 (negative) | 147
  AIS (positive) | 1
  AIS (negative) | 146
  Invasive malignancy (positive) | 0
  Invasive malignancy (negative) | 147
  Other | 56

6. Primary Outcome: Number of Subjects With Cervical Biopsy Results at Month 36
Description: as for outcome 4
Time Frame: At Month 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 88
Participants
  Negative | 31
  Only CIN1(positive) | 31
  Only CIN1(negative) | 57
  Only CIN2 (positive) | 6
  Only CIN2 (negative) | 82
  Only CIN3 (positive) | 3
  Only CIN3 (negative) | 85
  CIN1 and CIN2 (positive) | 0
  CIN1 and CIN2(negative) | 88
  CIN1 and CIN3(positive) | 0
  CIN1 and CIN3 (negative) | 88
  CIN2 and CIN3 (positive) | 0
  CIN2 and CIN3 (negative) | 88
  CIN1 and CIN2 and CIN3 (positive) | 0
  CIN1 and CIN2 and CIN3 (negative) | 88
  AIS (positive) | 0
  AIS (negative) | 88
  Invasive malignancy (positive) | 0
  Invasive malignancy (negative) | 88
  Other | 25

7. Primary Outcome: Number of Subjects With Cervical Biopsy Results at Month 48
Description: as for outcome 4
Time Frame: At Month 48
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 54
Participants
  Negative | 21
  Only CIN1(positive) | 15
  Only CIN1(negative) | 39
  Only CIN2 (positive) | 5
  Only CIN2 (negative) | 49
  Only CIN3 (positive) | 2
  Only CIN3 (negative) | 52
  CIN1 and CIN2 (positive) | 1
  CIN1 and CIN2(negative) | 53
  CIN1 and CIN3(positive) | 0
  CIN1 and CIN3 (negative) | 54
  CIN2 and CIN3 (positive) | 0
  CIN2 and CIN3 (negative) | 54
  CIN1 and CIN2 and CIN3 (positive) | 0
  CIN1 and CIN2 and CIN3 (negative) | 54
  AIS (positive) | 0
  AIS (negative) | 54
  Invasive malignancy (positive) | 0
  Invasive malignancy (negative) | 54
  Other | 11

8. Primary Outcome: Number of Subjects With Treatment Referrals by Treatment Type at Month 12
Description: If a high-grade lesion was detected, the subject was to be referred to treatment according to local medical practice. Any further management following local cervical therapy for cervical lesions was to be handled according to local medical practice within the local health care system. The subject's participation in the study concluded after treatment.
  The treatment types included the following: Loop excision of cervix, Loop cone of cervix, Cold knife cone of cervix, Laser excision, other.
Time Frame: At Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 392
Participants
  Treatment referral, Yes | 33
  Treatment referral, No | 359
  Loop excision of cervix, Yes: number analyzed (Participants) | 32
  Loop excision of cervix, Yes | 14
  Loop excision of cervix, No: number analyzed (Participants) | 32
  Loop excision of cervix, No | 18
  Loop cone of cervix, Yes: number analyzed (Participants) | 32
  Loop cone of cervix, Yes | 15
  Loop cone of cervix, No: number analyzed (Participants) | 32
  Loop cone of cervix, No | 17
  Cold knife cone of cervix, Yes: number analyzed (Participants) | 32
  Cold knife cone of cervix, Yes | 0
  Cold knife cone of cervix, No: number analyzed (Participants) | 32
  Cold knife cone of cervix, No | 32
  Laser excision, Yes: number analyzed (Participants) | 32
  Laser excision, Yes | 1
  Laser excision, No: number analyzed (Participants) | 32
  Laser excision, No | 31
  Other: number analyzed (Participants) | 32
  Other | 4

9. Primary Outcome: Number of Subjects With Treatment Referrals by Treatment Type at Month 24
Description: as for outcome 8
Time Frame: At Month 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 263
Participants
  Treatment referral, Yes | 19
  Treatment referral, No | 243
  Treatment referral, Missing | 1
  Loop excision of cervix, Yes: number analyzed (Participants) | 17
  Loop excision of cervix, Yes | 9
  Loop excision of cervix, No: number analyzed (Participants) | 17
  Loop excision of cervix, No | 8
  Loop cone of cervix, Yes: number analyzed (Participants) | 17
  Loop cone of cervix, Yes | 4
  Loop cone of cervix, No: number analyzed (Participants) | 17
  Loop cone of cervix, No | 13
  Cold knife cone of cervix, Yes: number analyzed (Participants) | 17
  Cold knife cone of cervix, Yes | 1
  Cold knife cone of cervix, No: number analyzed (Participants) | 17
  Cold knife cone of cervix, No | 16
  Laser excision, Yes: number analyzed (Participants) | 17
  Laser excision, Yes | 0
  Laser excision, No: number analyzed (Participants) | 17
  Laser excision, No | 17
  Other: number analyzed (Participants) | 17
  Other | 4

10. Primary Outcome: Number of Subjects With Treatment Referrals by Treatment Type at Month 36
Description: as for outcome 8
Time Frame: At Month 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 158
Participants
  Treatment referral, Yes | 13
  Treatment referral, No | 145
  Loop excision of cervix, Yes: number analyzed (Participants) | 10
  Loop excision of cervix, Yes | 4
  Loop excision of cervix, No: number analyzed (Participants) | 10
  Loop excision of cervix, No | 6
  Loop cone of cervix, Yes: number analyzed (Participants) | 10
  Loop cone of cervix, Yes | 4
  Loop cone of cervix, No: number analyzed (Participants) | 10
  Loop cone of cervix, No | 6
  Cold knife cone of cervix, Yes: number analyzed (Participants) | 10
  Cold knife cone of cervix, Yes | 0
  Cold knife cone of cervix, No: number analyzed (Participants) | 10
  Cold knife cone of cervix, No | 10
  Laser excision, Yes: number analyzed (Participants) | 10
  Laser excision, Yes | 0
  Laser excision, No: number analyzed (Participants) | 10
  Laser excision, No | 10
  Other: number analyzed (Participants) | 10
  Other | 2

11. Primary Outcome: Number of Subjects With Treatment Referrals by Treatment Type at Month 48
Description: as for outcome 8
Time Frame: At Month 48
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 96
Participants
  Treatment referral, Yes | 9
  Treatment referral, No \ | 87
  Loop excision of cervix, Yes: number analyzed (Participants) | 8
  Loop excision of cervix, Yes | 1
  Loop excision of cervix, No: number analyzed (Participants) | 8
  Loop excision of cervix, No | 7
  Loop cone of cervix, Yes: number analyzed (Participants) | 8
  Loop cone of cervix, Yes | 5
  Loop cone of cervix, No: number analyzed (Participants) | 8
  Loop cone of cervix, No | 3
  Cold knife cone of cervix, Yes: number analyzed (Participants) | 8
  Cold knife cone of cervix, Yes | 0
  Cold knife cone of cervix, No: number analyzed (Participants) | 8
  Cold knife cone of cervix, No | 8
  Laser excision, Yes: number analyzed (Participants) | 8
  Laser excision, Yes | 1
  Laser excision, No: number analyzed (Participants) | 8
  Laser excision, No | 7
  Other: number analyzed (Participants) | 8
  Other | 1

12. Primary Outcome: Number of Subjects With Adverse Events (AEs) or Serious Adverse Events (SAEs) Leading to Withdrawal
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: From Month 12 [i.e. 12 months after the last visit in HPV-008 (NCT00122681) primary study) up to Month 48 [i.e. 48 months after the last visit in HPV-008 (NCT00122681) primary study]
Population: The analysis was based on the Total HPV-052 cohort, which included subjects who had their symptom sheet completed and who at their last HPV-008 (NCT00122681) study visit displayed normal cervical cytology but tested positive for oncogenic HPV infection or were pregnant so that no cervical sample could be collected at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 2003
Participants | 216

13. Primary Outcome: Number of Subjects With Any Fatal SAEs, With Any SAEs Assessed as Possibly Related to Study Participation or to a Concurrent GSK Medication.
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-052 Study Subjects Group
Number analyzed (Participants) | 2003
Participants
  Subjects with fatal SAEs | 0
  Subjects with any related SAEs | 0
  Subjects with any SAEs due to concurrent GSK medic | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From Month 12 [i.e. 12 months after the last visit in HPV-008 (NCT00122681) primary study) up to Month 48 [i.e. 48 months after the last visit in HPV-008 (NCT00122681) primary study].
Description: Non-serious AEs were not collected in this study. Only fatal SAEs, SAEs related to study participation, SAEs related to a concurrent GSK medication and AEs and SAEs leading to withdrawal from the study were collected in this study.
Arm/Group | HPV-052 Study Subjects Group
All-Cause Mortality (participants affected / at risk) | 0/2003
Serious Adverse Events (participants affected / at risk) | 0/2003
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.